CLINICAL TRIAL: NCT00566306
Title: Influence of a New Polycationic Disinfectant on Clostridium Difficile Incidence and Environmental Colonisation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Soft Protector (Industry); The Finnish Funding Agency for Technology and Innovation (TEKES) (Other Government)
Responsible Party: Mari Kanerva, HUCH,Department of Medicine, Division of Infectious Diseases
Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 231109
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Clostridium Difficile
Keywords: Clostridium difficile; disinfectant
MeSH Terms: interventions — polyhexamethyleneguanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): PHMG will be introduced in three wards for hand hygiene and environmental disinfection in CDAD patients' rooms. The rooms for showers and toilets will be coated with biocide coating (PHMG) as well as bed frames in investigational wards.
  Interventions: Other: Polyhexamethyleneguanidine (PHMG)
- B (No Intervention): Three wards will be control wards and continue using alcohol based hand disinfectants and routine environmental cleaning and disinfection with quats/chloramines.

INTERVENTIONS:
Other: Polyhexamethyleneguanidine (PHMG) — 6 months in 3 experimental wards
  Other Names: Desisoft
  Arms: A

SUMMARY:
The aim of this study is to 1) test the efficacy of PHMG-based disinfectant against C. difficile spores, 2) test whether it reduces the incidence of C. difficile associated disease (CDAD) and 3) evaluate cost.

DETAILED DESCRIPTION:
Environmental disinfection has been proved to be efficient when controlling epidemics caused by C. difficile. In recent years its epidemiology has changed leading to increased morbidity and mortality in many countries. C. difficile infections are often difficult to treat and reinfections frequently occur. The major concern is a new strain of C. difficile, O27, which produce many times more spores than other types and spreads easily in institutions. Patients who have a C. difficile infection should be kept in contact isolation in hospitals and other institutions.

C. difficile is a spore forming bacteria which is resistant to some normally used disinfectants like alcohol and quats. Spores may remain viable for months in environment. Disinfectants currently in use, like chloramines and glutaralde-hyde, are risk both for workers and to environment because of their corrosive and irritating nature.

Polyhexamethyleneguanidine(PHMG) is a new disinfectant which is effective against microbes including bacteria and bacterial spores, viruses and fungi, safe to people handling it and friendly to environment and surfaces. It has been tested in the laboratory of Helsinki University according to many EN-standards to disinfectants. It can be used as a hand disinfectant, instrument disinfectant and surface disinfectant.

PHMG was introduced in three wards for hand hygiene and environmental disinfection in CDAD patients' rooms. The rooms for showers and toilets were coated with biocide coating (PHMG) as well as bed frames in investigational wards. Three wards were control wards and continued using alcohol based hand disinfectants and routine environmental cleaning and disinfection with quats/chloramines. After 6 month's intervention period, the incidence of CDAD cases were compared to that during the preceeding 10 months. Surveillance for environmental and HCWs´ hand contamination by C. difficile were performed by taking microbiological samples both from environmental sites and hands twice before intervention and then twice in month within intervention period.

ELIGIBILITY:
Inclusion Criteria: ( classified as a HCF-onset, HCF-associated CDAD )

* toxin or culture positive C difficile
* symptom onset more than 72 hours after admission to hospital
* symptom onset less than 4 weeks after discharge

Exclusion Criteria:

* recurrence of CDAD within 8 weeks
* symptom onset before admission to hospital or less than 72 hours after admission to hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Clinical: C. difficile infections on study wards. Microbiologic: C difficile colonization. | 2/07-5/08

SECONDARY OUTCOMES:
Economical: to evaluate cost of C difficile infection | 2/07-5/08

CONTACTS AND LOCATIONS:
Overall Officials: Mari Kanerva, MD,PhD, Principal Investigator — Helsinki University Central Hospital, Department of Medicine, Division of Infectious Diseases